CLINICAL TRIAL: NCT06475157
Title: Artificial Intelligence-enhanced Electrocardiogram Diagnoses and Predicts Future
Brief Title: Artificial Intelligence-enhanced Electrocardiogram Diagnoses and Predicts Future Regurgitant Valvular Heart Diseases
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AIECG_VHDP
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Electrocardiogram, Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group with progression of valvular heart diseases
  Interventions: Other: No intervention
- Patient group without progression of valvular heart diseases
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is applied.

SUMMARY:
This is a retrospective study to establish models for the prediction of future valvular heart diseases with artificial intelligence-enhanced electrocardiogram (ECG).

ELIGIBILITY:
Inclusion Criteria:

* Subjects that received ECG and echocardiography tests during a date frame.

Exclusion Criteria:

* Subjects who is younger than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An overall population.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Progression of valvular heart diseases | 15 years
  There would be echo records of subjectes of the study during follow-up. So for subjects with baseline none or mild valvular heart diseases, including mitral regurgitation, aortic regurgitation, and tricuspid regurgitation, there might be some with progression to moderate or severe valvular heart diseases, and some other without this progression. The primary outcome of the study would be the progression of valvular heart diseases from none or mild to moderateor severe, as assessed by echocardiography.

CONTACTS AND LOCATIONS:
Locations (2):
- 180 Fenglin Road, Shanghai, China
- Hammersmiths Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No